CLINICAL TRIAL: NCT00215917
Title: D-Serine Monotherapy for Schizophrenia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herzog Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: lichtenberg1CTIL
Record Dates: First submitted 2005-09-18; First posted 2005-09-22 (Estimated); Last update posted 2006-05-03 (Estimated); Status verified 2006-05

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; NMDA; D-serine
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Drug: D-serine 2100 mg daily

SUMMARY:
N-methyl-D-aspartate receptor (NMDAR) agonist, added to classical or atypical antipsychotic medication, has reduced negative, depressive, and cognitive symptomatology. We will be investigating the effect of D-serine, (DSR), a selective and potent NMDAR agonist, as monotherapy for treatment resistant schizophrenics.

40 subjects on stable doses of risperidone will be randomized under double-blind conditions into a treatment group, which will receive D-serine 2100 mg, or a control group, which will continue to receive risperidone. Treatment will continue for 14 weeks.

Symptoms and side effects will be rated biweekly with the CGI, PANSS, BPRS, SAS, AIMS, and UKU. Before and after the trial subjects will undergo neuropsychological assessments. Baseline and post-trial levels of amino acids relevant to glutamatergic neurotransmission (glutamate, glutamine, aspartate, glycine, serine, alanine) will be assessed.

The primary outcome measures of the study will be the PANSS total scores and the positive and negative symptom cluster scores.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV criteria for chronic schizophrenia
2. Treatment resistant
3. aged 18-70
4. Two months on stable risperidone dose
5. PANSS positive symptom cluster score >20
6. PANSS negative symptom cluster score >22

Exclusion Criteria:

1. Substance abuse
2. Concurrent DSM IV axis I disorder
3. Serious medical disorder
4. Concurrent drug therapy that can obscure the effect of risperidone or DSR.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40

CONTACTS AND LOCATIONS:
Overall Officials: Pesach Lichtenberg, M.D., Principal Investigator — Herzog Hospital, and Hadassah Medical School--the Hebrew University of Jerusalem, Israel
Locations (1):
- Herzog Hospital, Department of Psychiatry, Jerusalem, Israel